CLINICAL TRIAL: NCT00003296
Title: Phase II Study of TLC D-99 for Hepatobiliary Carcinomas
Brief Title: Liposomal Doxorubicin in Treating Patients With Liver or Bile Duct Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brown University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066230; BRUOG-HB-71; NCI-V98-1408
Record Dates: First submitted 1999-11-01; First posted 2004-07-08 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2000-09

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; localized gallbladder cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; localized extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; adult primary hepatocellular carcinoma; cholangiocarcinoma of the gallbladder; cholangiocarcinoma of the extrahepatic bile duct; adult primary cholangiocellular carcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Filgrastim

INTERVENTIONS:
Biological: filgrastim
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of liposomal doxorubicin in treating patients with liver or bile duct cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and toxicity of doxorubicin HCl liposome in patients with carcinomas of the liver and bile ducts.

OUTLINE: Patients receive doxorubicin HCl liposome IV over 15 minutes every 21 days. Filgrastim (G-CSF) is administered subcutaneously starting on day 2 and continuing for 10-14 days. Disease is restaged after every 3 courses. Treatment continues in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for the first year, and then every 6 months thereafter.

PROJECTED ACCRUAL: There will be 17-26 evaluable patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed carcinoma of the liver or bile ducts including hepatocellular carcinoma, cholangiocarcinoma, and gallbladder cancer Measurable or evaluable disease by CT scan (ascites, pleural effusions, and bone metastases are not considered evaluable)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 3 mg/dL No severe cirrhosis Renal: Creatinine no greater than 3.0 mg/dL Cardiovascular: Left ventricular cardiac ejection fraction at least 45% Other: No allergy to egg or egg products Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior doxorubicin At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — Brown University
Locations (2):
- United States (2):
  - New England Medical Center Hospital, Boston, Massachusetts
  - Brown University Oncology Group, Providence, Rhode Island